CLINICAL TRIAL: NCT00971100
Title: A Randomized, Single-blind, Dose-Ranging Study to Evaluate Immunogenicity, Safety and Tolerability of Different Formulations of Adjuvanted and Non Adjuvanted Cell-derived, Inactivated Novel Swine Origin A/H1N1 Monovalent Subunit Influenza Virus Vaccine in Healthy Subjects From 6 Months to 17 Years of Age
Brief Title: Immunogenicity, Safety and Tolerability of Two Doses of Adjuvanted and Non-adjuvanted Swine Origin A/H1N1 Monovalent Influenza Vaccine in Healthy Subjects From 6 Months to 17 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V110_04; 2009-013640-37 (EudraCT Number)
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2011-10

CONDITIONS: Pandemic Influenza
Keywords: Pandemic influenza; Vaccine

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- low dose of antigen + low dose of adjuvant (Experimental)
  Interventions: Biological: Monovalent A/H1N1 influenza vaccine
- high dose of antigen + high dose of adjuvant (Experimental)
  Interventions: Biological: Monovalent A/H1N1 influenza vaccine
- high dose of antigen (Experimental)
  Interventions: Biological: Monovalent A/H1N1 influenza vaccine

INTERVENTIONS:
Biological: Monovalent A/H1N1 influenza vaccine — This trial will be performed at multiple study sites in a population of healthy children and adolescent. Subjects will be randomized to receive 2 IM injections of low dose of antigen & adjuvant, or high dose of antigen & adjuvant, or high dose of antigen, according to the study groups.

SUMMARY:
The present study, randomized, single-blind, dose-ranging, multicenter study, will evaluate immunogenicity, safety and tolerability of two doses of adjuvanted and not-adjuvanted new swine-origin influenza A/H1N1 virus monovalent subunit vaccine in healthy children and adolescents. A booster dose will be administered 12 months after the first vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 6 months of age to 17 years of age on the day of enrollment;
2. Subject's parents or legal guardians who have given written consent and the subjects has given assent consent, if applicable;
3. Individuals in good health;
4. Subjects, subject's parents or legal guardians that are able to comply with all study procedures;
5. Willingness to allow for serum samples to be stored beyond the study period, for potential additional future testing to better characterize immune response.

Exclusion Criteria:

1. Subject's parents or legal guardians who are not able to comprehend and to follow all required study procedures;
2. Individuals with history or any illness that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study;
3. Individuals with any serious chronic or progressive disease according to judgment of the investigator;
4. History of any anaphylaxis, serious vaccine reactions to any excipients and to eggs (including ovalbumin) and chicken protein;
5. Individuals who have had adjuvanted influenza vaccine or documented confirmed or suspected influenza disease within 3 months prior to Day 1.
6. Receipt of another investigational agent within 4 weeks prior to enrollment or before completion of the safety follow-up period in this or in another study, unwilling to refuse a participation in another clinical study through the end of this study;
7. Individuals who receive any other vaccine 4 weeks prior to enrolment in this study or who are planning to receive any vaccine within four weeks from the study vaccines; the only exception being plain seasonal influenza vaccines which are allowed until one week prior to and after one week study vaccinations;
8. Individuals who have received blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation in the past 12 weeks;
9. Individuals with axillary temperature ≥ 38.0 degrees Celsius within 3 days of intended study vaccination;
10. Known or suspected alteration of immune function;
11. History of progressive or severe neurologic disorder;
12. Surgery planned during the study period that in the Investigator's opinion would interfere with the study visits schedule;
13. If female, of childbearing potential, and has not used any of the "acceptable contraceptive methods" for at least 2 months prior to study entry;
14. Females who are pregnant or nursing (breastfeeding) mothers, or females of childbearing potential do not plan to use acceptable birth control measures during the first 3 weeks after vaccination;
15. Members of research staff or their relatives.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 752 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To identify the preferred vaccine formulation dosage (antigen & adjuvant) and schedule (one or two administrations) of the H1N1sw monovalent vaccine in children and adolescents | 43 days after first vaccination

SECONDARY OUTCOMES:
To evaluate immunogenicity against A/California H1N1sw strain after booster dose of egg-derived seasonal trivalent, MF59 adjuvanted vaccine Fluad, recommended for 2010/2011 season, administered 12 months after primary course according to CHMP criteria. | 3 weeks after booster vaccination

CONTACTS AND LOCATIONS:
Locations (3):
- Gent, Antwerpen, Belgium
- Santo Domingo, Dominican Republic
- Wurzburg, Fulda, Neumunster, Balve, Leipzig, Rostock, Detmold, Mainz, Germany

REFERENCES:
- [Result] Knuf M, Leroux-Roels G, Rumke H, Rivera L, Pedotti P, Arora AK, Lattanzi M, Kieninger D, Cioppa GD. Immunogenicity and safety of cell-derived MF59(R)-adjuvanted A/H1N1 influenza vaccine for children. Hum Vaccin Immunother. 2015;11(2):358-76. doi: 10.4161/21645515.2014.987014. PMID 25621884